CLINICAL TRIAL: NCT03793998
Title: Catheter Ablation of Arrhythmias With High Density Mapping System in the Real World Practice. The CHARISMA Study
Brief Title: Catheter Ablation of Arrhythmias With High Density Mapping System in the Real World Practice.
Acronym: CHARISMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Pugliese Ciaccio (Other)
Responsible Party: Principal Investigator, Giampiero Maglia, Head of Electrophysiology and Cardiac Pacing, Azienda Ospedaliera Pugliese Ciaccio
Other Study IDs: Protocollo n. 89 (17/04/2018)
Record Dates: First submitted 2018-11-29; First posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Cardiac Arrhythmias
Keywords: Cardiac Catheter Ablation; Cardiac Arrhythmias; Mapping System
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

SUMMARY:
The CHARISMA study is a non-randomized, multicenter, prospective study in which consecutive patients indicated for arrhythmia will be enrolled.

Patients can be treated with any market released catheter for ablation and diagnostic examination. The decision to perform the ablation will be made based on clinical evaluation of the investigators according to their clinical practice. The study does not require specific surgical techniques. The study has been designed to describe the Italian clinical practice in relation to the ablation approach of different kind of arrhythmias. In particular, the investigators will analyze the percentage of acute and long-term success in clinical practice, predictors of arrhythmias recurrence and they will describe the methods for the validation of ablation success, the techniques adopted, and the patient management approaches in the participating centers

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible for ablation procedure of atrial and ventricular arrhythmia;
* Patients who are able to sign an authorization to use and disclose health information and capable of providing informed consent.
* Patients who are willing and capable to attend scheduled follow-up visits at the clinical investigational center for at least 12 months

Exclusion Criteria:

* Patients who are currently enrolled in another clinical study that would directly interfere with the clinical practice of the investigational center

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients, clinically indicated for arrhythmias ablation, will be enrolled after signing an informed consent form and an authorization to use and disclose health information
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with arrhythmia recurrences | 12 months
  The primary outcome measure of this study is to estimate, after 12-months from the procedure, the percentage of patients with documented arrhythmia recurrences, recognized with the registration of at least 30 seconds of the same arrhythmias with 24h Holter ECG

SECONDARY OUTCOMES:
The percentage of acute procedural success of arrhythmias ablation | within 30 minutes after ablation procedure
  This secondary outcome measures the percentage of acute procedural success. The acute success of the arrhythmias ablation is verified by; the completion of the necessary ablation application(s), the validation of ablation through appropriate technique(s) and, when applicable, the termination of the primary arrhythmia.
Baseline patient's characteristic (clinical history and drug therapy) for subjects undergoing catheter ablation | within 30 minutes after ablation procedure
  This secondary outcome measures the baseline patient's characteristics (clinical history and drug therapy) as potential predictors of acute success
Rate of new onset of different arrhythmias (from the primary one) | 12 months
  This secondary outcome measures the rate of new onset of any kind of different arrhythmia (from the primary one) related to the primary ablation procedure
Primary arrhythmia recurrences and association with the baseline patient's characteristics (clinical history and drug therapy) | 36 months
  This secondary outcome measure of this study is to evaluate baseline patient's characteristics as potential predictors of primary arrhythmia recurrences, that will be evaluated at 12 months and 36 months follow up
Overall procedure time | Intraoperative
  This secondary outcome measures the radiofrequency delivery time, the total ablation time, the fluoroscopy time
Rate of the adverse events associated with the primary ablation procedure | 12 months
  This secondary outcome measures the rate of the adverse events that occurs during the procedure and after 12 months
Estimate costs related to the use of health care resources | 60 months
  This secondary outcome measures the resource consumption and the associated costs in term of ablation procedures, follow-up, management of complication and health care resources utilization

CONTACTS AND LOCATIONS:
Overall Officials: Giampiero Maglia, MD, Principal Investigator — Azienda Ospedaliera Pugliese Ciaccio
Locations (1):
- Azienda Ospedaliera Pugliese-Ciaccio, Catanzaro, Italy

REFERENCES:
- [Derived] Mantovan R, Bianchi S, Pelargonio G, Solimene F, Malacrida M, Carbone A, Anselmino M, Gallucci M, Segreti L, Galeazzi M, Bianco D, Giomi A, Mirizzi G, Rossi L, Zingarini G, Calvanese R, Allocca G, Ducceschi V, Dell'Era G, Bisignani A, Scacciavillani R, Schillaci V, Rivetti L, Bulian F. Ultra High-Density Mapping and Ablation of Localized Micro-Reentrant Tachycardias: Insight From the CHARISMA Registry. J Cardiovasc Electrophysiol. 2025 Apr;36(4):794-806. doi: 10.1111/jce.16563. Epub 2025 Jan 30. PMID 39888109
- [Derived] Schiavone M, Bianchi S, Malacrida M, Fassini G, Ricciolino R, Pecora D, Pelargonio G, Iacopino S, Ducceschi V, Maggio R, Bianchini L, La Greca C, Rossi P, Bencardino G, Moltrasio M, Di Belardino N, Pepi P, Rossi L, Santagostino M, Tondo C, De Simone A. Novel cryoballoon technology for atrial fibrillation ablation: Impact of pulmonary vein variant anatomy, cooling characteristics, and 1-year outcome from the CHARISMA registry. Heart Rhythm. 2025 May;22(5):1134-1141. doi: 10.1016/j.hrthm.2024.08.040. Epub 2024 Aug 22. PMID 39181485
- [Derived] Solimene F, Maggio R, De Sanctis V, Escande W, Malacrida M, Stabile G, Zakine C, Champ-Rigot L, Anselmino M, Ferraro A, Mantica M, Zucchelli G, Dell'Era G, Mascia G, Ricci Maga R, Pandozi C, Rossi P, Scaglione M, Zingarini G, Garnier F, Loricchio ML, Pelargonio G, Lepillier A. Contact-force local impedance algorithm to guide effective pulmonary vein isolation in AF patients: 1-year outcome from an international multicenter clinical setting. J Interv Card Electrophysiol. 2024 Dec;67(9):2137-2146. doi: 10.1007/s10840-024-01849-0. Epub 2024 Jul 8. PMID 38972960
- [Derived] Bianchi S, De Simone A, Iacopino S, Fassini G, Malacrida M, Rossi P, Stabile G, Petretta A, Tundo F, Cauti FM, Iuliano S, Filannino P, Moltrasio M, Morlacchi Bonfanti M, Pelargonio G, Pecora D, Ferraro A, Tondo C. Pulmonary vein isolation by means of a novel cryoballoon technology in paroxysmal atrial fibrillation patients: 1-year outcome from a large Italian multicenter clinical registry. Pacing Clin Electrophysiol. 2023 Nov;46(11):1302-1309. doi: 10.1111/pace.14839. Epub 2023 Oct 17. PMID 37846769
- [Derived] Lepillier A, Maggio R, De Sanctis V, Malacrida M, Stabile G, Zakine C, Champ-Rigot L, Anselmino M, Segreti L, Dell'Era G, Garnier F, Mascia G, Pandozi C, Dello Russo A, Scaglione M, Cosaro G, Ferraro A, Paziaud O, Maglia G, Solimene F. Insight into contact force local impedance technology for predicting effective pulmonary vein isolation. Front Cardiovasc Med. 2023 Jul 5;10:1169037. doi: 10.3389/fcvm.2023.1169037. eCollection 2023. PMID 37476572
- [Derived] Schillaci V, Arestia A, Maddaluno F, Shopova G, Agresta A, Salito A, Stabile G, Marano G, Bottaro G, Malacrida M, Solimene F. Combining contact force and local impedance to treat idiopathic premature ventricular contractions from the outflow tracts: impact of ablation strategy on outcomes. J Interv Card Electrophysiol. 2023 Dec;66(9):2011-2020. doi: 10.1007/s10840-023-01528-6. Epub 2023 Mar 24. PMID 36964415
- [Derived] Spera F, Narducci ML, Bencardino G, Perna F, Bisignani A, Pinnacchio G, Tondo C, Maggio R, Stabile G, Iacopino S, Tundo F, Ferraro A, De Simone A, Malacrida M, Pintus F, Crea F, Pelargonio G. Ultra-high-resolution assessment of lesion extension after cryoballoon ablation for pulmonary vein isolation. Front Cardiovasc Med. 2022 Nov 9;9:985182. doi: 10.3389/fcvm.2022.985182. eCollection 2022. PMID 36439999
- [Derived] Solimene F, Stabile G, Segreti L, Malacrida M, Schillaci V, Rossi P, Bongiorni MG, Shopova G, Cauti FM, Zucchelli G, Arestia A, Bianchi S, Di Cori A, Maddaluno F, De Simone A, Garcia-Bolao I. Targeted ablation of residual pulmonary vein potentials in atrial fibrillation ablation through ultra-high-density mapping: Insights from the CHARISMA registry. J Cardiovasc Electrophysiol. 2022 Jul;33(7):1414-1424. doi: 10.1111/jce.15527. Epub 2022 Jun 1. PMID 35524404
- [Derived] Ducceschi V, Zingarini G, Nigro G, Brasca FMA, Malacrida M, Carbone A, Lavalle C, Maglia G, Infusino T, Aloia A, Nicolis D, Auricchio C, Uccello A, Notaristefano F, Rago A, Botto GL, Esposito L. Optimized radiofrequency lesions through local impedance guidance for effective CTI ablation in right atrial flutter. Pacing Clin Electrophysiol. 2022 May;45(5):612-618. doi: 10.1111/pace.14482. Epub 2022 Apr 22. PMID 35383979
- [Derived] Solimene F, De Sanctis V, Maggio R, Malacrida M, Segreti L, Anselmino M, Schillaci V, Mantica M, Scaglione M, Dello Russo A, Cauti FM, Zingarini G, Pandozi C, Cavaiani M, Ferraro A, Maglia G, Stabile G. When local impedance meets contact force: preliminary experience from the CHARISMA registry. J Interv Card Electrophysiol. 2022 Apr;63(3):749-758. doi: 10.1007/s10840-022-01163-7. Epub 2022 Mar 24. PMID 35322330
- [Derived] Iacopino S, Stabile G, Fassini G, De Simone A, Petretta A, Moltrasio M, La Rocca V, Placentino F, Riva S, Pesce F, Rossi P, Pelargonio G, Iuliano A, Tundo F, Colella J, Tondo C. Key characteristics for effective acute pulmonary vein isolation when using a novel cryoballoon technology: insights from the CHARISMA registry. J Interv Card Electrophysiol. 2022 Sep;64(3):641-648. doi: 10.1007/s10840-021-01063-2. Epub 2021 Dec 2. PMID 34853986
- [Derived] Pandozi C, Lavalle C, Bongiorni MG, Catalano A, Pelargonio G, Russo M, Piro A, Carbone A, Narducci ML, Galeazzi M, Ficili S, Piccolo F, Maddaluno F, Malacrida M, Colivicchi F, Segreti L. High-density mapping of Koch's triangle during sinus rhythm and typical AV nodal reentrant tachycardia: new insight. J Interv Card Electrophysiol. 2021 Sep;61(3):487-497. doi: 10.1007/s10840-020-00841-8. Epub 2020 Aug 6. PMID 32766944